CLINICAL TRIAL: NCT06237530
Title: Exploring Visceral Body Scan, Somatosensory Body Scan, and External Meditation
Brief Title: Interoception and Body Scan
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rosa M. Baños Rivera, Full Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2569173
Record Dates: First submitted 2023-12-04; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Healthy
Keywords: body scan; interoception; interoceptive; mindfulness; somatosensory

STUDY DESIGN:
Intervention Model Description: The investigators tested two different versions of the body scan (meditation practice), one focused on visceral signals -visceral body scan (VBS)- and the other on somatosensory signals -somatosensory body scan (SBS)- in comparison to an exteroceptive, non-body focused, control condition -external control meditation (ECM)-. To do so, an online approach was conducted, as it has been proved to be an effective strategy, while being more widely accessible and reducing costs and time.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Visceral Body Scan (VBS) (Experimental): The VBS consisted of a mindfulness exercise designed to bring awareness to visceral sensations in the cardiac, respiratory, gastrointestinal, and urinary systems. These physiological systems were chosen because most of the paradigms developed in the literature to assess interoception focus on them (Khalsa et al., and they are widely recognized in the literature as interoceptive senses (Nord & Garfinkel, 2022)
  Interventions: Behavioral: Visceral body scan (VBS)
- Somatosensory body scan (SBS) (Active Comparator): The SBS consisted of a mindfulness exercise designed to bring awareness to tactile (e.g., itching) and musculoskeletal (e.g. g., tension) sensations in different parts of the body, namely, the head and neck, back, arms, and legs. Body scan exercises typically focus on these types of bodily cues (in addition to breathing) (Williams, 2010).
  Interventions: Behavioral: Somatosensory body scan (SBS)
- External control meditation (ECM) (Sham Comparator): The ECM consisted of a mindfulness exercise designed to bring awareness to external stimuli, including sounds and visual properties of the environment
  Interventions: Behavioral: External control meditation (ECM)

INTERVENTIONS:
Behavioral: Visceral body scan (VBS) — The VBS consisted of a mindfulness exercise designed to bring awareness to visceral sensations in the cardiac, respiratory, gastrointestinal, and urinary systems. These physiological systems were chosen because most of the paradigms developed in the literature to assess interoception focus on them (Khalsa et al., and they are widely recognized in the literature as interoceptive senses (Nord & Garfinkel, 2022)
  Other Names: Interoceptive body scan; Interoceptive meditation practice
  Arms: Visceral Body Scan (VBS)
Behavioral: Somatosensory body scan (SBS) — The SBS consisted of a mindfulness exercise designed to bring awareness to tactile (e.g., itching) and musculoskeletal (e.g. g., tension) sensations in different parts of the body, namely, the head and neck, back, arms, and legs. Body scan exercises typically focus on these types of bodily cues (in addition to breathing) (Williams, 2010).
  Other Names: Exteroceptive body scan; Somatosensory meditation practice
  Arms: Somatosensory body scan (SBS)
Behavioral: External control meditation (ECM) — The ECM consisted of a mindfulness exercise designed to bring awareness to external stimuli, including sounds and visual properties of the environment.
  Other Names: Non-body meditation practice; Visual and auditory mindfulness exercise
  Arms: External control meditation (ECM)

SUMMARY:
Body scan meditation has been assumed to be an interoceptive intervention, and the evidence for its effects on interoceptive processes is unclear. Although this mindfulness based exercise typically involves focusing on some interoceptive signals such as breath, it also involves other bodily cues, such as somatosensory cues. The present study aimed to (1) investigate the feasibility of three online delivered mindfulness practices that differ in the signals targeted: visceral body scan (VBS), somatosensory body scan (SBS), and external (non body) meditation (ECM), and (2) gain insight into the potentially different effects of these interventions on interoceptive and other psychological outcomes in order to inform future full scale randomized controlled trials (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* being Spanish or English speakers
* Ability to use a computer or smartphone
* Daily access to computer or smartphone with an Internet connection

Exclusion Criteria:

* Being diagnosed with a severe psychiatric disorder (e.g., substance abuse, eating disorder, psychotic disorder)
* Severe visual or auditory difficulties that cannot be corrected with glasses or auditory aids
* Having a medical condition that prevents participation in this study
* Changes in psychotropic medication during the study
* Having been exposed to any extremely traumatic event that is being re-experienced or interfering during the last month
* Body image-related difficulties as indicated by scores above 3 on the Body Image as Source of Shame questionnaire.
* Regular meditation practice in the current moment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Adherence assessed by completed intervention sessions | Through study completion, a total of 7 days
  Percentage of completed daily sessions during the 7-day intervention
Meditation-related adverse effects assessed by a self-report questionnaire | Immediately post-intervention
  Meditation-Related Adverse Effect Scale - Mindfulness-Based Program. It includes 11 dichotomic items (yes/no questions), so scores ranges from 0 to 11, with higher scores indicating more adverse effects
Acceptability assessed by a satisfaction questionnaire | Immediately post-intervention
  Treatment Satisfaction Scale. It includes 5 items rated on Likert-point scale ranging from 0 to 10. Thus, total scores range from 0 to 50, with higher scores indicating greater acceptability of the intervention
Self-reported quality of the mindfulness practice | Immediately post-intervention
  Practice Quality-Mindfulness. It consists of 6 items rated on a visual analogue scale ranging from 0 to 100, with higher scores reflecting a higher level of practice quality.

SECONDARY OUTCOMES:
Adaptive interoceptive sensibility style assessed by a questionnaire | Immediately pre-intervention and immediately post-intervention
  Multidimensional Assessment of Interoceptive Awareness-2. It consists of 37 items rated on a 6-point Likert scale, with higher values indicating a more adaptive and healthier interoceptive sensibility style (healthier approach to internal bodily signals).
Sensitivity and attention to interoceptive signals assessed by a questionnaire | Immediately pre-intervention and immediately post-intervention
  Interoceptive Sensitivity and Attention Questionnaire. It consists of 17 items rated on a 5-point Likert scale, ranging from 1 (totally disagree) to 5 (totally agree). Higher scores reflect greater sensitivity to bodily sensations
Perceived Body Boundaries in bodily self-awareness assessed by a VAS | Immediately pre-intervention and immediately post-intervention
  Perceived Body Boundaries Scale. It is visual analogue scale that depicts seven human bodies, ranging from almost imperceptible at the left pole (labeled "my body boundaries are almost imperceptible") to extremely salient at the right pole (labeled my body boundaries are extremely salient"). Scores can range from 0 to 15.5, with higher scores indicating greater salience in perceiving body boundaries.
Spatial Frame of Reference in bodily self-awareness assessed by a VAS | Immediately pre-intervention and immediately post-intervention
  Spatial Frame of Reference Continuum. It is a visual analogue scale depicting five concentric circles surrounding the outline of a human figure, and individuals are asked to indicate how far they feel that their self extends beyond their physical body. Scores range from 1 to 6, with higher scores reflecting a more allocentric (vs. egocentric) frame of reference.
Mindfulness trait assessed by a self-report questionnaire | Immediately pre-intervention and immediately post-intervention
  Short form of the Five Facet Mindfulness Questionnaire. It is a 15-item instrument that measures the tendency to be mindful in daily life. Items are rated on a 5-point Likert scale, from 1 (never or very rarely true) to 5 (very often or always true). It includes the following dimensions: observing, describing, acting with awareness, non judging internal experience, and non reactivity to internal experience. Higher scores indicate higher levels of the corresponding mindfulness dimension.
Alexithymia assessed by a self-report questionnaire | Immediately pre-intervention and immediately post-intervention
  The Perth Alexithymia Questionnaire Questionnaire-Short Form. It includes 7 items rated on a 7-point Likert scale (1=strongly disagree; 7=strongly agree), with higher scores indicating higher levels of alexithymia
Negative emotion regulation assessed by a self-report questionnaire | Immediately pre-intervention and immediately post-intervention
  Short-form version of the Difficulties in Emotion Regulation Scale. It is an 18 item questionnaire that measures the degree of difficulty in regulating emotions. Items are rated on a 5 point Likert scale, ranging from 1 (almost never) to 5 almost always). It includes the following dimensions: (1) lack of emotional awareness of one's own emotions; (2) self reported difficulty in completing tasks and concentrating in the presence of negative emotions; (3) limited access to regulatory strategies that the in dividual perceives as effective; (4) nonacceptance of negative emotional states; (5) self reported difficulty in controlling one's behavior in the presence of negative emotional states, and (6) lack of emotional clarity, i.e., limited knowledge and clarity about one's emotional states. Higher scores indicate higher difficulties in regulating emotions.
Positive emotion regulation assessed by a self-report questionnaire | Immediately pre-intervention and immediately post-intervention
  Responses to Positive Affect Questionnaire. It is a 16 item questionnaire that measures responses to positive moods, including dampening (i.e., thoughts that are likely to dampen positive emotional states), self focused positive rumination (i.e., rumination on aspects of the self and the pursuit of goals relevant to the self), and emotion focused positive rumination (i.e., rumination on positive mood). Items are rated on a 4 point Likert scale, ranging from 1 almost never ) to 4 almost always ), with higher scores reflecting a greater use of such strategy.
Depressive symptomatology assessed by a self-report questionnaire | Immediately pre-intervention and immediately post-intervention
  Patient Health Questionnaire-9. It consists of 9 items, which are rated on a 4-point Likert scale, ranging from 0 (never) to 4 (almost every day). Higher scores indicate greater severity of depressive symptoms.
Qualitative feedback assessed by several open-ended questions | Immediately pre-intervention and immediately post-intervention
  Ad-hoc open-ended questions: ended questions: (1) "Do you think that participating in this study has helped you learn something or become aware of something? If so, what did you learn?"; (2) Do you think that doing the meditation practice has helped you improve anything? If so, what benefits have you noticed noticed?"; (3) Does this practice make sense to you, and why? "; (4) Please describe the sensations, thoughts and/or feelings you have had while doing the meditation practice "; (5) What difficulties have you found when doing the meditation practice?"; (6) What did you like most about the meditation practice? And what did you like the least?", and (7) What do you think is the objective or hypothesis of the study?".

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Baños, PhD, Principal Investigator — Univeristy of Valencia
Locations (1):
- Faculty of Psychology and Speech Therapy, University of Valencia, Valencia, Valencia, Spain